CLINICAL TRIAL: NCT05720429
Title: Evaluation of the Usefulness and Feasibility of a Psychoeducational Intervention to Prevent the Negative Psychological Impact of the COVID-19 Pandemic on Primary Health Care Professionals
Brief Title: A Psychoeducational Intervention to Prevent the Psychological Impact of COVID-19 Pandemic in Primary Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Fundació Galatea (Unknown); Institut Català de la Salut (Other); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Enric Aragonès, Senior Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SLT021/21/000028; 4R22/033 (Other: IDIAPJGol)
Record Dates: First submitted 2023-01-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Issue; Burnout, Professional
Keywords: mental health; health personnel; primary health care; COVID-19 pandemic; psychological support
MeSH Terms: conditions — Burnout, Professional; Psychological Well-Being; COVID-19

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pragmatic study in a real clinical practice environment with a design before after with mixed quantitative-qualitative methodology. The intervention will be carried out in a decentralized way through the primary care centres of the Catalan Health Institute (over 250). All of the groups are supposed to receive the same intervention, although the diverse range of experiences will be described and measured as part of the program's implementation feasibility evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary care workers (Experimental): Primary care health personnel who will voluntarily join the psychoeducational program of their center.
  All professional profiles working in primary care centers are eligible (ie primary care nurses, physiotherapists, family doctors, pediatricians, dentists, administrative staff, etc.). Groups of 10-15 people. Several groups can be established in the same center if the demand is high enough.
  Interventions: Other: Psychoeducational program

INTERVENTIONS:
Other: Psychoeducational program — A psychoeducational program consisting of 11 one-hour sessions, with a weekly or biweekly frequency, each one regarding specific tools and skills to promote emotional well-being, self-care, and the ability to deal with stressful situations. They are conducted by community psychologists, who will give a brief theoretical introduction and then conduct practical group exercises that apply the concepts introduced. Every session ends with a relaxation exercise and some habits that the participants can incorporate into their daily life.
  Session Index: (1) Emotional management;(2) Thought management; (3) Stress management; (4) Communication skills, active listening, and empathy; (5) Self-care; (6) Individual/group self-esteem; (7) Anxiety/coping with panic. Mindfulness; (8) Activating motivation; (9) Problem-Solving; (10) Positive psychology and emotional intelligence; (11) Emotional expression through art.
  Other Names: Programa Ventilació Emocional

SUMMARY:
The goal of this quasi-experimental pragmatic study is to design, implement and evaluate a psychoeducational group intervention aimed at preventing the negative consequences of the COVID-19 pandemic on the psychological wellbeing and mental health of primary care healthcare workers.

The experience will be carried out in real clinical practice conditions and our purpose is to evaluate it not only in terms of clinical effectiveness but, especially, the terms of feasibility, usefulness, and possibility of this intervention being integrated into the usual practice in primary care centers.

There will be two types of participation and a mixed quantitative-qualitative methodology. On one hand, the healthcare workers that will receive the intervention and participate in the study by responding to various before and after online surveys with standardized scales. On the other hand, the community psychologists in charge of implementing the intervention, having received guidelines and training, will help gather the participants' data and will provide their perceptions, assessments, and opinions on the program through other questionnaires. After the intervention, a selection of both healthcare workers and psychologists will participate in qualitative in-depth, or group interviews to explore the nuances of their perceptions of the program.

The results will allow the investigators to know the usefulness and effectiveness of the intervention and, above all, to model and improve its design and implementation strategy, and promote its generalization beyond the framework of this project.

DETAILED DESCRIPTION:
The COVID-19 pandemic has constituted an extraordinarily stressful situation for healthcare professionals and has generated an impact in the form of psychological distress and the appearance of various mental health disorders. In this context, it is necessary to provide these professionals with strategies and skills to be able to manage stressful situations and prevent or minimize their negative impact.

The investigators hypothesize that the implementation of a psychoeducational group intervention framed in the Primary Care Emotional Well-Being Program (Department of Health) may be feasible, useful, and effective to prevent harmful psychological effects and increase the emotional well-being of healthcare professionals in the context of the pandemic.

General objective: To analyze the implementation of a psychological group intervention for the promotion/prevention of mental health and the improvement of the psychological distress of primary care professionals in relation to the COVID-19 pandemic.

Specific objectives:

* Measure the clinical effects of the intervention in terms of psychological symptoms, burnout, and health-related quality of life.
* Identify predictor factors concerning the clinical effects of the intervention
* Identify different profiles of professionals based on their clinical response
* To explore from a qualitative perspective the perceptions and assessments of the healthcare professionals who receive it and the community psychologists who apply it regarding barriers, facilitators, and proposals for improving the program and the implementation strategy.
* Modeling/perfecting/individualizing the intervention

Design: Quasi-experimental pragmatic study in a real clinical practice environment with a design before-after with mixed quantitative-qualitative methodology.

Intervention: A psychoeducational program aimed at all professional roles of primary care workers, designed by an expert group and implemented by the community psychologists from the Primary Care Emotional Well-Being Program. It consists of eleven sessions about different tools and skills to promote emotional well-being and improve the ability to deal with stressful situations, developed with an eminently practical approach.

The strategy for the implementation and deployment of the intervention includes facilitators such as an intervention manual and an online training course for the psychologists who will apply it.

Measurements:

1. On the procedure of implementation: a set of quantitatively measurable indicators that cover different aspects of quality and performance of the implementation process (number of editions of the intervention, number of participants, adherence of participants, etc.).
2. On the clinical effect on participants: through standardized questionnaires that participants must fill out autonomously. A prospective evaluation of the main outcome variables (quality of working life, burnout, psychological state) will be carried out with basal evaluation points, before starting the intervention, at the end of the intervention, at 3 and 6 months.

Sub-study of qualitative methodology. Design: Study with a phenomenological approach to know the perceptions and assessments of the participants regarding the applied psychoeducational intervention. Collection of information: individual in-depth interviews and online group interviews, aimed at (a) health workers participating in psychoeducational groups, and (b) community psychologists who apply the intervention.

Scope. This experience will be carried out in the primary care centers of the Catalan Health Institute. Over 18 months, editions of psychoeducational activity will be carried out in a decentralized way.

The results will allow the investigators to know the usefulness and effectiveness of the intervention and, above all, to model and improve its design and implementation strategy, and promote its generalization beyond the framework of this project.

ELIGIBILITY:
Inclusion Criteria:

* Workers of Primary Care Healthcare Centers, from the Catalan Health Institute and other functionally dependent centers. Any professional profile.
* Participants in group psychoeducational programs organized by community psychologists in their centers.

Exclusion Criteria:

* Being currently diagnosticated with a severe mental health disorder.
* Being in a litigation process due to inability to work due to a psychological disorder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ProQOL Health Care Workers version | Change from baseline (before the intervention) to immediately after the intervention
  Professional Quality of Life Scale, Health Care Workers version. A questionnaire with 30 items that reflect health workers' feelings and perceptions concerning their work. The items are answered on a Likert scale according to frequency, from 1 ("never") to 5 points ("always").
  The following dimensions are evaluated: (1) Compassion satisfaction, which measures the satisfaction of being able to work well; (2) Perceived support; (3) Burnout; (4) Secondary traumatic stress, related to secondary exposure to stressful events in work; and (5) Moral distress, which reflects the conflict of facing difficult choices or in contradiction with personal values. The dimensions of compassion satisfaction and perceived support are considered health worker strengths, and burnout, traumatic stress, and moral distress are vulnerabilities.
ProQOL Health Care Workers version | Change from baseline (before the intervention) to 3 months following the intervention
  Professional Quality of Life Scale, Health Care Workers version. A questionnaire with 30 items that reflect health workers' feelings and perceptions concerning their work. The items are answered on a Likert scale according to frequency, from 1 ("never") to 5 points ("always").
  The following dimensions are evaluated: (1) Compassion satisfaction, which measures the satisfaction of being able to work well; (2) Perceived support; (3) Burnout; (4) Secondary traumatic stress, related to secondary exposure to stressful events in work; and (5) Moral distress, which reflects the conflict of facing difficult choices or in contradiction with personal values. The dimensions of compassion satisfaction and perceived support are considered health worker strengths, and burnout, traumatic stress, and moral distress are vulnerabilities.
ProQOL Health Care Workers version | Change from baseline (before the intervention) to 6 months following the intervention
  Professional Quality of Life Scale, Health Care Workers version. A questionnaire with 30 items that reflect health workers' feelings and perceptions concerning their work. The items are answered on a Likert scale according to frequency, from 1 ("never") to 5 points ("always").
  The following dimensions are evaluated: (1) Compassion satisfaction, which measures the satisfaction of being able to work well; (2) Perceived support; (3) Burnout; (4) Secondary traumatic stress, related to secondary exposure to stressful events in work; and (5) Moral distress, which reflects the conflict of facing difficult choices or in contradiction with personal values. The dimensions of compassion satisfaction and perceived support are considered health worker strengths, and burnout, traumatic stress, and moral distress are vulnerabilities.
CD-RISC10 | Change from baseline (before the intervention) to immediately after the intervention
  10-item Connor-Davidson Resilience Scale. A unidimensional self-reported scale consisting of 10 items measuring resilience. Respondents rate items on a 5-point Likert scale (0-4).
CD-RISC10 | Change from baseline (before the intervention) to 3 months following the intervention
  10-item Connor-Davidson Resilience Scale. A unidimensional self-reported scale consisting of 10 items measuring resilience. Respondents rate items on a 5-point Likert scale (0-4).
CD-RISC10 | Change from baseline (before the intervention) to 6 months following the intervention
  10-item Connor-Davidson Resilience Scale. A unidimensional self-reported scale consisting of 10 items measuring resilience. Respondents rate items on a 5-point Likert scale (0-4).
DASS-21 | Change from baseline (before the intervention) to immediately after the intervention
  Depression Anxiety and Stress Scale, 21 items. The DASS-21 contains three scales that assess the presence of symptoms or indicators of depression, anxiety, and stress. Each scale has seven items that are rated on a Likert scale from 0 points ("never happens to me") to 3 points ("almost always or always happens to me").
DASS-21 | Change from baseline (before the intervention) to 3 months following the intervention
  Depression Anxiety and Stress Scale, 21 items. The DASS-21 contains three scales that assess the presence of symptoms or indicators of depression, anxiety, and stress. Each scale has seven items that are rated on a Likert scale from 0 points ("never happens to me") to 3 points ("almost always or always happens to me").
DASS-21 | Change from baseline (before the intervention) to 6 months following the intervention
  Depression Anxiety and Stress Scale, 21 items. The DASS-21 contains three scales that assess the presence of symptoms or indicators of depression, anxiety, and stress. Each scale has seven items that are rated on a Likert scale from 0 points ("never happens to me") to 3 points ("almost always or always happens to me").

OTHER OUTCOMES:
Qualitative research: facilitators | Up to six months after the intervention completion
  Facilitators of program implementation assessed using qualitative research methods
Qualitative research: barriers | Up to six months after the intervention completion
  Barriers of program implementation assessed using qualitative research methods
Qualitative research: proposals for improvement | Up to six months after the intervention completion
  Proposals for improvement of the psychoeducational program assessed using qualitative research methods

CONTACTS AND LOCATIONS:
Overall Officials: Enric Aragonès Benaiges, MD, PhD, Principal Investigator — IDIAPJgol; Josep Basora Gallisà, MD, PhD, Study Chair — IDIAPJgol; Francisco M Martín Luján, MD, PhD, Study Chair — IDIAPJgol; Anna Berenguera Ossó, DrPH, Study Chair — IDIAPJgol; Ariadna Mas Casals, MD, Study Chair — Institut Català de la Salut; Sara Rodoreda Noguerola, MD, Study Chair — Institut Català de la Salut; Antoni Calvo López, Study Chair — Fundació Galatea, Fundació Privada; Concepción Rambla Vidal, MD, Study Chair — IDIAPJgol; Meritxell Guitart Peces, Study Chair — ICS; Eva García Cots, Study Chair — ICS
Locations (1):
- Institut Universitari d'Investigació en Atenció Primària IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llor C, Moragas A. [Coronavirus and primary care]. Aten Primaria. 2020 May;52(5):294-296. doi: 10.1016/j.aprim.2020.03.002. Epub 2020 Apr 6. No abstract available. Spanish. PMID 32284192
- [Background] Garcia-Alegria J, Gomez-Huelgas R. COVID-19 disease: the hospital of the future is already here. Rev Clin Esp (Barc). 2020 Oct;220(7):439-441. doi: 10.1016/j.rce.2020.05.010. Epub 2020 Jun 3. No abstract available. PMID 32560916
- [Background] Barba R. [Healthcare management during COVID-19 pandemia.]. Arch Esp Urol. 2020 Jun;73(5):330-335. Spanish. PMID 32538801
- [Background] Alonso J, Vilagut G, Mortier P, Ferrer M, Alayo I, Aragon-Pena A, Aragones E, Campos M, Cura-Gonzalez ID, Emparanza JI, Espuga M, Forjaz MJ, Gonzalez-Pinto A, Haro JM, Lopez-Fresnena N, Salazar ADM, Molina JD, Orti-Lucas RM, Parellada M, Pelayo-Teran JM, Perez-Zapata A, Pijoan JI, Plana N, Puig MT, Rius C, Rodriguez-Blazquez C, Sanz F, Serra C, Kessler RC, Bruffaerts R, Vieta E, Perez-Sola V; MINDCOVID Working group. Mental health impact of the first wave of COVID-19 pandemic on Spanish healthcare workers: A large cross-sectional survey. Rev Psiquiatr Salud Ment (Engl Ed). 2021 Apr-Jun;14(2):90-105. doi: 10.1016/j.rpsm.2020.12.001. Epub 2020 Dec 10. PMID 33309957
- [Background] Martinez-Lopez JA, Lazaro-Perez C, Gomez-Galan J, Fernandez-Martinez MDM. Psychological Impact of COVID-19 Emergency on Health Professionals: Burnout Incidence at the Most Critical Period in Spain. J Clin Med. 2020 Sep 20;9(9):3029. doi: 10.3390/jcm9093029. PMID 32962258
- [Background] Aragones E, Fernandez-San-Martin M, Rodriguez-Barragan M, Martin-Lujan F, Solanes M, Berenguera A, Siso A, Basora J. Gender differences in GPs' strategies for coping with the stress of the COVID-19 pandemic in Catalonia: A cross-sectional study. Eur J Gen Pract. 2023 Dec;29(2):2155135. doi: 10.1080/13814788.2022.2155135. Epub 2022 Dec 19. PMID 36533663
- [Background] Maunder RG, Lancee WJ, Balderson KE, Bennett JP, Borgundvaag B, Evans S, Fernandes CM, Goldbloom DS, Gupta M, Hunter JJ, McGillis Hall L, Nagle LM, Pain C, Peczeniuk SS, Raymond G, Read N, Rourke SB, Steinberg RJ, Stewart TE, VanDeVelde-Coke S, Veldhorst GG, Wasylenki DA. Long-term psychological and occupational effects of providing hospital healthcare during SARS outbreak. Emerg Infect Dis. 2006 Dec;12(12):1924-32. doi: 10.3201/eid1212.060584. PMID 17326946
- [Background] Pollock A, Campbell P, Cheyne J, Cowie J, Davis B, McCallum J, McGill K, Elders A, Hagen S, McClurg D, Torrens C, Maxwell M. Interventions to support the resilience and mental health of frontline health and social care professionals during and after a disease outbreak, epidemic or pandemic: a mixed methods systematic review. Cochrane Database Syst Rev. 2020 Nov 5;11(11):CD013779. doi: 10.1002/14651858.CD013779. PMID 33150970
- [Background] Jimenez-Gimenez M, Sanchez-Escribano A, Figuero-Oltra MM, Bonilla-Rodriguez J, Garcia-Sanchez B, Rojo-Tejero N, Sanchez-Gonzalez MA, Munoz-Lorenzo L. Taking Care of Those Who Care: Attending Psychological Needs of Health Workers in a Hospital in Madrid (Spain) During the COVID-19 Pandemic. Curr Psychiatry Rep. 2021 Jun 19;23(7):44. doi: 10.1007/s11920-021-01253-9. PMID 34152465
- [Background] Galiana L, Arena F, Oliver A, Sanso N, Benito E. Compassion Satisfaction, Compassion Fatigue, and Burnout in Spain and Brazil: ProQOL Validation and Cross-cultural Diagnosis. J Pain Symptom Manage. 2017 Mar;53(3):598-604. doi: 10.1016/j.jpainsymman.2016.09.014. Epub 2017 Jan 3. PMID 28062348
- [Background] Stetler CB, Damschroder LJ, Helfrich CD, Hagedorn HJ. A Guide for applying a revised version of the PARIHS framework for implementation. Implement Sci. 2011 Aug 30;6:99. doi: 10.1186/1748-5908-6-99. PMID 21878092
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Novy DM, Stanley MA, Averill P, Daza P. Psychometric comparability of English- and Spanish-language measures of anxiety and related affective symptoms. Psychol Assess. 2001 Sep;13(3):347-55. doi: 10.1037//1040-3590.13.3.347. PMID 11556271
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Derived] Aragones E, Rodoreda S, Guitart M, Garcia E, Berenguera A, Martin F, Rambla C, Aragones G, Calvo A, Mas A, Basora J. Study protocol: assessment of the usefulness and practicability of a psychoeducational intervention to prevent the negative psychological impact of the COVID-19 pandemic on primary care health workers. BMC Prim Care. 2023 Nov 4;24(1):231. doi: 10.1186/s12875-023-02187-2. PMID 37925394
- See also: Intervention Manual — https://drive.google.com/file/d/1lz-9nC1AlN7AyW1c4jtA531fkRkQGHPt/view?usp=share_link
- See also: Online course for training implementers. user: ventilacioemocional password: convidat123 — https://campus.idiapjgol.org/course/view.php?id=48
- See also: Online course videos — https://www.youtube.com/playlist?list=PLcUX3bp5a6GTacx-I7onAb3GKtDasJwZc
- See also: Procedure for RBEC implementers — https://docs.google.com/document/d/1S1B5HMFK2Y87VCRJPHEC8_yQAT9qxYQ10G9uxJyl7d0/edit#heading=h.dkwk82s5y2zh